CLINICAL TRIAL: NCT03890471
Title: Telephone Intervention to Increase Patient Preparedness and Satisfaction Trial (TIPPS): A Randomized Control Trial Evaluating the Effect of Preoperative Telephone Calls on Patient Preparedness and Satisfaction in Urogynecologic Surgery
Brief Title: Telephone Intervention to Increase Patient Preparedness and Satisfaction Trial (TIPPS): A Randomized Control Trial
Acronym: TIPPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Gabriela Halder, Principle Investigator, FPMRS Fellow, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2018120057
Record Dates: First submitted 2019-03-11; First posted 2019-03-26 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Prolapse; Stress Urinary Incontinence
MeSH Terms: conditions — Prolapse; Urinary Incontinence, Stress

STUDY DESIGN:
Intervention Model Description: We will conduct a randomized controlled trial comparing a provider-initiated preoperative telephone call plus usual clinic counseling to usual clinic counseling alone in women planning pelvic reconstructive surgery for SUI and/or POP.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preoperative telephone call (Experimental): Patients will receive routine preoperative counseling in the clinic plus a provider initiated telephone call 3 days before surgery.
  Interventions: Behavioral: Preoperative telephone call three days before surgery
- No preoperative telephone call (No Intervention): Patients will receive routine preoperative counseling in the clinic.

INTERVENTIONS:
Behavioral: Preoperative telephone call three days before surgery — Patients will receive a provider-initiated telephone call three days before surgery. In order to standardize counseling across providers, each provider will use a telephone script addressing the following components: Purpose of the surgery, alternatives to the surgery, surgical benefits, surgical risk (such as infection, bleeding, injury to other organ systems), potential surgical complications (such as mesh erosion, voiding dysfunction, urinary retention requiring indwelling catheter), bowel complaints (such as nausea, vomiting, constipation, diarrhea), and postoperative expectations (such as Foley management, pain management, activity restrictions, and diet. The following ERAS-specific components will be incorporated into the counseling: management of chronic medical conditions, cessation of alcohol and tobacco, and daily exercise until surgery. Questions from patients and total counseling time will be recorded.
  Arms: Preoperative telephone call

SUMMARY:
Surgical preparedness improves patient satisfaction and perioperative outcomes. In urogynecology, interventions to increase preoperative patient preparedness have not been adequately studied. Our objective is to evaluate the ability of preoperative provider-initiated telephone calls to increase patient preparedness for surgery. The investigators will conduct a randomized control trial comparing surgical preparedness between provider-initiated telephone call three days before surgery plus usual preoperative counseling versus usual preoperative counseling alone among women planning to undergo pelvic reconstructive surgery as measured by the Preoperative Patient Questionnaire (PPQ) and the Modified Preparedness for Colorectal Cancer Surgery Questionnaire (Modified PCSQ). Surgical satisfaction, perioperative outcomes, and medical costs will be also be compared between the two groups. Our hypothesis is that preoperative telephone calls will result in improved surgical preparedness. This novel approach in preoperative counseling has the potential to positively impact perioperative patient care.

The investigators will also conduct an ancillary qualitative study of sexually active women undergoing pelvic reconstructive surgery who are enrolled in the randomized control trial. This work will aim to describe the patient experience, concerns, and the quality of the first sexual encounter following surgery. This ancillary study will lay the foundation for future investigations into how to better counsel patients and discuss sexual activity after surgical repair.

DETAILED DESCRIPTION:
Increased surgical preparedness is linked to improved surgical satisfaction and patient-reported outcomes. Interventions that increase preparedness for surgery are needed. The impact of a provider-initiated preoperative telephone call on surgical preparedness is unknown. The objectives of this study are to compare patient preparedness between women who receive a preoperative provider-initiated telephone call plus the usual preoperative counseling in the clinic versus usual preoperative counseling alone. The investigators hypothesize that a provider initiated preoperative telephone call will increase surgical preparedness and satisfaction, as well as improve perioperative outcomes. The investigators will test our working hypothesis by using the approach of randomizing patients undergoing surgery for SUI and/or POP to either a provider-initiated telephone call three days before surgery plus usual preoperative counseling or usual preoperative counseling alone. The rationale for this aim is that successful completion of the proposed research will contribute a missing, fundamental element to our understanding of preoperative counseling. It is our expectation that a preoperative telephone call three days before surgery will result in improved surgical preparedness. Such a finding would be of importance because it would provide evidence to support a novel method in preoperative counseling that positively impacts patient care.

Patients enrolled in the ancillary sexual function study will be scheduled for one-on-one telephone interview 2-4 months after surgery. Major themes of the interviews will be used to better describe the patient experience of return to sexual activity after surgery.

The investigators are also planning on performing a cost analysis. A provider-initiated telephone call before surgery requires the allocation of new resources that may result in additional perioperative costs. However, if telephone calls improve perioperative outcomes, an overall decrease in perioperative costs may be observed due to a decrease in direct and non-direct costs. Direct costs are attributable to the use of a health care intervention or illness and can be further classified in medical and non-medical costs. Medical care costs include emergency room visits, hospital admissions, unplanned clinic visits, clinic telephone calls. Non-medical costs include transportation, gas, and parking. Indirect costs include lost wages for the patient or caregiver. The objective of aspect of the study is to determine the difference in cost-effectiveness between women who receive a provider-initiated telephone call 3 days before surgery plus the usual preoperative counseling in the clinic versus the usual preoperative counseling alone from the patient and societal perspectives. The investigators hypothesize that preoperative telephone calls will be more cost-effective for both patients and society. The investigators will test our working hypothesis by using the approach of resource costing method. It is our expectation that preoperative telephone calls will improve perioperative outcomes resulting in overall cost to both the patient and society that will compensate for the additional perioperative costs associated with a telephone call before surgery.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Speak and read English: Only English-speaking women will be allowed to participate because the questionnaires used in the study are validated only in English and Swedish; they are not validated in other languages.
* Planned surgery for pelvic organ prolapse and/or stress urinary incontinence

Exclusion Criteria:

* Less than 18 years of age
* Do not read or speak English
* Unable to participate in a telephone call (dementia, hard of hearing, deaf)
* Scheduled for surgery in 3 days or less

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2019-06-05 (Actual); Primary Completion 2020-05-11 (Actual); Study Completion 2020-05-11 (Actual)

PRIMARY OUTCOMES:
Surgical preparedness | Baseline
  Patient Preparedness Questionnaire, Modified Preparedness for Colorectal Cancer Surgery Questionnaire

SECONDARY OUTCOMES:
Surgical satisfaction | Will be measured at postoperative visit 4-8 weeks after surgery.
  Decision Regret Scale and Satisfaction with Decision Scale, Scale of 1-5, Scoring consists of reversing the scores of the 2 negatively phrased items, then taking the mean of the 5 items (range, 1-5).
Patient-reported outcomes | Will be measured at baseline and at the postoperative visit 4-8 weeks after surgery.
  Pelvic Floor Distress Inventory - 20
Cost-effectiveness | Will be measured at baseline and at the postoperative visit 4-8 weeks after surgery.
  The European Quality of Life-5 Dimensions

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Rogers, MD, Principal Investigator — Tenured Processor, Department of Women's Health at UT Austin
Locations (2):
- United States (2):
  - Seton Midtown Medical Tower, Austin, Texas
  - Pelvic Floor Integrated Practice Unit at the University of Texas Health Austin, Austin, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Halder GE, Guo F, Harvie H, White AB, Caldwell L, Giles DL, Bilagi D, Rogers RG. Cost Effectiveness of Additional Preoperative Telephone Call to Increase Surgical Preparedness: Analysis of a Randomized Clinical Trial. Int Urogynecol J. 2024 Mar;35(3):527-536. doi: 10.1007/s00192-023-05719-7. Epub 2024 Jan 8. PMID 38189853